CLINICAL TRIAL: NCT02896062
Title: Development and Evaluation of a Sleep-coaching Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Heidi Danker-Hopfe, Head of Competence Center of Sleep Medicine, Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: M/SAKE/EA002
Record Dates: First submitted 2016-08-31; First posted 2016-09-12 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group (Experimental): In the treatment phase subjects receive a sleep-coaching
  Interventions: Behavioral: sleep-coaching
- Waiting group control (Active Comparator): The waiting group receives the treatment after a waiting period of up to 6 weeks
  Interventions: Behavioral: sleep-coaching

INTERVENTIONS:
Behavioral: sleep-coaching — Sleep-coaching with elements of cognitive behavioral therapy for insomnia and general information about sleep

SUMMARY:
In the present study, a 4-week sleep coaching program is developed and evaluated in members of the German armed Forces. The aim of the program is to provide an efficient tool to prevent sleep disorders, and to improve mild sleep disorders, with a special focus on insomnia.

DETAILED DESCRIPTION:
In the present study, a sleep-coaching program for small groups of a maximum of eight participants is developed. The program is comprised of four different sessions and is provided to member of the German armed forces. One session lasts approximately 1.5 hours and sessions are applied on a weekly basis. Each session deals with a different topic, addressing all major categories of sleep disorders (insomnia, hypersomnia, circadian rhythm disorders, sleep-related breathing disorders) and teaching ways of self-help and information on when to seek medical treatment. The program is evaluated by a cross-over study design with treatment and waiting control groups. After the treatment group has finished the course, the waiting group attends the sleep coaching session. All subjects fill in sleep logs and several questionnaires prior to (t0) and after the treatment group has finished the sleep coaching (t1), after the waiting group has finished the course (t2), and in a 3-month follow-up session (t3). Furthermore, sleep is recorded according to the AASM-standard criteria for two consecutive nights each at the time-points t0, t1, and t2. Subjective and objective sleep quality will be compared across the time-points, and between groups. In total, at least 48 participants are included in study.

ELIGIBILITY:
Inclusion Criteria:

* subjectively impaired sleep quality
* member of the German armed forces

Exclusion Criteria:

* subjects with a clinically relevant psychiatric decease
* not able to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
subjective sleep quality assessed by PSQI | 5 months
  PSQI total score

SECONDARY OUTCOMES:
objective sleep quality assessed by PSG | 2 months
  sleep efficiency

CONTACTS AND LOCATIONS:
Locations (1):
- Charité - University Medicine Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sauter C, Kowalski JT, Stein M, Rottger S, Danker-Hopfe H. Effects of a Workplace-Based Sleep Health Program on Sleep in Members of the German Armed Forces. J Clin Sleep Med. 2019 Mar 15;15(3):417-429. doi: 10.5664/jcsm.7666. PMID 30853042